CLINICAL TRIAL: NCT06425250
Title: Campylobacter Spp. Bone and Joint Infection: a Retrospective Cohort Study
Acronym: Campylo-BJI
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL23_5284
Record Dates: First submitted 2024-05-17; First posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Campylobacter Infections
Keywords: Management; Risk factors; Campylobacter spp.
MeSH Terms: conditions — Campylobacter Infections | interventions — Therapeutics; Risk Factors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Management, progression and risk factors for failure of BJI caused by Campylobacter spp.: Adult patients treated for prosthetic joint infection caused by Campylobacter spp. between 01/01/2013 and 12/31/2022
  Interventions: Other: Management, progression and risk factors for failure of BJI caused by Campylobacter spp.; Other: Description of the evolution and risk factors for failure of osteoarticular infections caused by Campylobacter spp.

INTERVENTIONS:
Other: Management, progression and risk factors for failure of BJI caused by Campylobacter spp. — Description of demographic data (sex, age), comorbidities (ASA and Charlson scores), orthopedic and septic history, and surgical and medical management (antibiotic therapy)
Other: Description of the evolution and risk factors for failure of osteoarticular infections caused by Campylobacter spp. — Failure of treatment: defined according to a composite criterion bringing together
  * persistence of the infection under treatment, and/or
  * recurrence of the infection after stopping antibiotic therapy, and/or
  * need for surgical revision for septic reasons more than 5 days after initial treatment, and/or
  * superinfection, and/or
  * definitive explantation of the material, and/or
  * decision for suppressive antibiotic therapy, and/or
  * amputation, and/or
  * death linked to infection

SUMMARY:
Campylobacter bacteria, a Gram-negative bacillus commensal in the digestive tract of many animals and mainly responsible for human infections with digestive origins, has been little studied in the field of osteoarticular infections (OAI). Campylobacter spp. are, however, well described, mainly for C. fetus, and pose a dual therapeutic problem: i) a capacity for persistence due to the capacity of most strains to form biofilm; and ii) potential resistance to many antibiotics. The management of IOA caused by Campylobacter spp. is not codified, and is based on small series of cases reported in the literature.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years
* Osteoarticular infection (whatever its type), mono or polymicrobial with Campylobacter spp., diagnosed between 01/01/2013 and 12/31/2022:
* Septic arthritis: compatible clinical signs + joint fluid sample positive in culture and/or PCR positive for Campylobacter
* Spondylodiscitis: clinical signs and MRI compatible + blood cultures and/or disco-vertebral biopsy puncture positive in culture and/or PCR positive for Campylobacter
* Osteitis/osteomyelitis: compatible clinico-radiological picture + bone sample (biopsy or intraoperative sample) positive in culture and/or positive PCR for Campylobacter
* Infection on joint prosthesis or osteosynthesis equipment: documented Campylobacter infection and meeting the definition of probable or confirmed JIBS infections
* Patient who was informed and did not object to participating in the study

Exclusion Criteria:

-

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients treated for prosthetic joint infection caused by Campylobacter spp. between 01/01/2013 and 12/31/2022
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Outcome of Campylobacter spp. BJI, measured as the proportion of treatment failure. | Outcome will be measure at 1 year. For patients lost of follow-up or followed-up less than a year, the date of last visit will be used for survival curve analysis .
  Treatment failure will be defined as: i) infection persistence under appropriate antimicrobial therapy; ii) infection relapse; iii) need for unplaned surgery; iv) superinfection and/or v) infection-related death

CONTACTS AND LOCATIONS:
Locations (1):
- Service des maladies infectieuses et tropicales - Hôpital de la Croix-Rousse, Lyon, France